CLINICAL TRIAL: NCT01600638
Title: Non-Invasive Reduction of Fat in the Flanks of Patients With Sharp Body Curvature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZA12-005
Record Dates: First submitted 2012-04-16; First posted 2012-05-17 (Estimated); Results first posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Body Fat Disorder
Keywords: Lipolysis; Cryolipolysis; Fat Reduction
MeSH Terms: interventions — Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Zeltiq System Treatment Group (Experimental): Individuals with sharp flank curvatures were treated on one (1) flank with the Zeltiq CoolSculpting System and the CoolCurve+ applicator at protocol-defined temperatures and durations.
  Interventions: Device: The Zeltiq System

INTERVENTIONS:
Device: The Zeltiq System — Non-invasive cooling is applied to the treatment area with a defined cooling rate and duration.
  Other Names: Cryolipolysis; Lipolysis

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the ZELTIQ System and the CoolCurve+ applicator for non-invasive fat reduction in flanks for a patient population with sharp body curvature.

DETAILED DESCRIPTION:
The Zeltiq System with the CoolCurve+ applicator will be evaluated for safety and effectiveness in subjects with subcutaneous fat on the flanks and who have sharp body curvatures. The curvature of interest is typical of individuals who are relatively thin with a small body frame.

ELIGIBILITY:
Inclusion Criteria

* Male or female subjects > 18 years of age and < 65 years of age.
* Subject has clearly visible fat on the flanks, which in the investigator's opinion, may benefit from the treatment.
* Subject has not had weight change exceeding 10 pounds in the preceding month.
* Subject with body mass index (BMI) up to 29. BMI is defined as weight in pounds multiplied by 703 divided by the square of the height in inches.
* Subject with sharp flank curvature that fits well with the CoolCurve+ applicator.
* Subject agrees to maintain his/her weight (i.e., within 5 pounds) by not making any major changes in their diet or lifestyle during the course of the study.
* Subject has read and signed a written informed consent form.

Exclusion Criteria

* Subject has had a surgical procedure(s) in the area of intended treatment.
* Subject has had an invasive fat reduction procedure (e.g., liposuction, abdominoplasty, mesotherapy) in the area of intended treatment.
* Subject has had a non-invasive fat reduction and/or body contouring procedure in the area of intended treatment within the past 12 months.
* Subject needs to administer, or has a known history of subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
* Subject has a known history of cryoglobulinemia, cold urticaria, or paroxysmal cold hemoglobinuria.
* Subject has a known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
* Subject has a history of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
* Subject is taking or has taken diet pills or supplements within the past month.
* Subject has any dermatological conditions, such as moderate to excessive skin laxity, or scars in the location of the treatment sites that may interfere with the treatment or evaluation (stretch marks is not an exclusion).
* Subject has an active implanted device such as a pacemaker, defibrillator, or drug delivery system
* Subject is pregnant or intending to become pregnant during the study period (in the next 5 months).
* Subject is lactating or has been lactating in the past 6 months.
* Subject is unable or unwilling to comply with the study requirements.
* Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
* Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-03-29 (Actual); Primary Completion 2012-08-29 (Actual); Study Completion 2013-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bachelor, MD, Principal Investigator — Innovation Research Center
Locations (1):
- Innovation Research Center, Pleasanton, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Zeltiq System Treatment Group: All subjects treated with the Zeltiq System are included in the treatment arm.
  The Zeltiq System: Non-invasive cooling is applied to the treatment area with a defined cooling rate and duration.
Period: Overall Study
Arm/Group | Zeltiq System Treatment Group
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Zeltiq System Treatment Group
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 37.9 [21.9 to 54.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 13
  Caucasian | 9
  Hispanic | 2
  Middle Eastern | 1
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Safety of the Zeltiq System for Non-invasive Fat Reduction in Subjects With Greater Flank Curvature.
Description: Safety will be assessed by determination of the number of Unanticipated Adverse Device Effects (UADE) at the 8-week and 16-week post-treatment visits.
Time Frame: 8 weeks and 16 weeks post final treatment
Population: All subjects treated with the Zeltiq System were included in the analysis population.
Measure: Number; unit: UADEs
Arm/Group | Zeltiq System Treatment Group
Number analyzed (Participants) | 25
UADEs
  UADE reported at 8 weeks | 0
  UADE reported at 16 weeks | 0

2. Primary Outcome: Change in Fat Layer Thickness When Compared to Untreated Control
Description: Change in the fat layer thickness will be calculated by comparison of pre-treatment and 16 week post-treatment ultrasound measurements taken in the area treated with the device, and in the contralateral untreated control area. The Sponsor's standardized techniques for obtaining ultrasound imaging will be used. Overall fat layer thickness changes were normalized for each subject by subtracting the change in the untreated control from the change in treated area to remove the influence of weight variations. Results indicate the mm of fat layer reduction in the treated area.
Time Frame: 16 weeks post final treatment
Population: All subjects treated with the Zeltiq System were included in the analysis population.
Measure: Mean (Standard Error); unit: mm
Arm/Group | Zeltiq System Treatment Group
Number analyzed (Participants) | 25
mm | -1.3 (0.27)
Statistical Analysis 1: Comparison: Zeltiq System Treatment Group; Test type: Other; Mean Difference (Net) = -1.3, Standard Error of Mean 0.27

3. Secondary Outcome: Proportion of Pre-treatment Images Correctly Identified
Description: Change in the treated vs. untreated areas will be assessed by observation of changes in surface contour and/or fat volume by an independent photo review of pre-treatment and post-treatment images of the treated areas. Reviewers will be practicing dermatologists or plastic surgeons. All reviewers will be blinded to post-treatment vs. baseline untreated area. The order in which images will be presented will be randomized; for each subject placement of the baseline, pre-treatment image will be randomized for each pair of subject images. Reviewers will be asked to select the baseline photos for each subject photo series and record selections on a data collection form. Results reflect the proportion of correctly identified images.
Time Frame: 16 weeks post final treatment
Population: All eligible subjects treated with the Zeltiq System and who maintained weight within protocol requirements were included in the analysis population. Paired photos of each subject were reviewed by 3 independent reviewers to properly identify pre-treatment images.
Measure: Count of Units; unit: photos
Units Other Than Participants: photos
Arm/Group | Zeltiq System Treatment Group
Number analyzed (Participants) | 23
Number analyzed (photos) | 69
photos | 54
Statistical Analysis 1: Comparison: Zeltiq System Treatment Group; Test type: Other; sucess proportion = .7823, 95% CI 2-sided [0.614 to 0.951]

4. Secondary Outcome: Subject Satisfaction Questionnaire
Description: Subject satisfaction with the Zeltiq procedure as determined by the results of a subjects satisfaction questionnaire at the 16 week follow up visit.
Time Frame: 16 weeks post final treatment
Measure: Number; unit: percentage of participants
Arm/Group | Zeltiq System Treatment Group
Number analyzed (Participants) | 25
percentage of participants
  Procedure was somewhat to very comfortable | 80
  Feel a difference in treated area | 36
  Somewhat to very visible fat reduction | 40
  Overall effect was more than or about was expected | 80
  Overall satisfaction with procedure | 92
  Would have area re-treated again | 88
  Would repeat procedure | 44
  Would have additional areas treated | 16
  Would recommend procedure to a friend | 100

5. Secondary Outcome: Additional Safety Evaluation
Description: The number of device or procedure-related adverse events will be evaluated. The investigator determines if the Zeltiq CoolSculpting System (device) or the treatment (procedure) are related to all reported adverse events.
Time Frame: Enrollment though 16 weeks post final treatment
Population: All subjects treated with the Zeltiq System were included in the analysis population.
Measure: Number; unit: Device/ procedure-related AE's
Arm/Group | Zeltiq System Treatment Group
Number analyzed (Participants) | 25
Device/ procedure-related AE's | 3

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time of enrollment through the 16 week post-final follow-up visit.
Description: An adverse event is defined as any untoward medical occurrence in a subject, regardless of whether the event is related to the device. Averse Device Effect is defined as any sign, symptom, or disease in a study subject that occurs during the course of a clinical trial that is determined by the investigator to have a causal relationship or possible causal relationship with the device under investigation.
Arm/Group | Zeltiq System Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 3/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zeltiq System Treatment Group (N=25)
Prolonged numbness (Skin and subcutaneous tissue disorders) | 2 (2) — Both events considered related to the investigational device and were mild in severity.
Kidney infection (Infections and infestations) | 1 (1) — Not related to device or procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No